CLINICAL TRIAL: NCT05652465
Title: An Open Trial of Transcranial Magnetic Stimulation for Youth With Treatment-Resistant Major Depressive Disorder
Brief Title: Transcranial Magnetic Stimulation for Youth With Treatment-Resistant Major Depressive Disorder
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: We have not been able to enroll subjects. We will re-evaluate recruitment approach.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000776; 000776-M
Record Dates: First submitted 2022-12-14; First posted 2022-12-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06-30

CONDITIONS: Major Depressive Disorder
Keywords: TMS; Emotion; Magnetic Resonance Imaging; Brain Stimulation; CBT
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Active (Experimental): TMS
  Interventions: Device: Intermittent theta burst repetitive transcranial magnetic stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta burst repetitive transcranial magnetic stimulation (iTBS) — Device described in protocol

SUMMARY:
Background:

Major depressive disorder (MDD) is one of the most impairing medical conditions in the world. Medication and some kinds of talk therapy are standard treatments for teens with MDD, but these do not work well for everyone. Transcranial magnetic stimulation (TMS) has been approved to treat MDD in adults. TMS might help adolescents, too.

Objective:

To test TMS combined with cognitive behavioral therapy (CBT) in teens with MDD.

Eligibility:

People aged 13 to 17 years with MDD that has not responded to treatment.

Design:

Participants will be screened. They will have a physical exam and psychiatric evaluation. They will have an MRI scan and a test of their heart function. They will enroll in 2 NIH protocols (01-M-0254 and 18-M-0037).

For 2 to 6 weeks, participants will have weekly CBT, a kind of talk therapy. They will taper off of their psychiatric medicines.

For 2 weeks, participants will come to the clinic every weekday. They will receive 3 or 4 sessions of TMS on each of those days. A wire coil will be held on their scalp. A brief electrical current in the coil creates a magnetic pulse that affects brain activity. They will receive 30 TMS pulses in 10-second bursts; these will be repeated 60 times in each 15-minute session. Participants may hear a click and feel a pulling sensation under the coil. They may feel their muscles twitch. Each day, they will have tests of concentration, thinking, and memory. Some may have a 3rd week of TMS.

Participants will remain in the study for 5 more weeks. They will begin taking their medications again.

DETAILED DESCRIPTION:
Study Description:

This is a safety and pilot efficacy study of open, neuronavigated intermittent theta burst stimulation (iTBS), a form of repetitive transcranial magnetic stimulation (rTMS) in medication-free youth with treatment-resistant major depression. The hypothesis is that intermittent theta burst TMS is a safe and potentially effective treatment for treatment-resistant major depression in adolescents.

Objectives:

The study has two objectives: 1) To evaluate safety, feasibility, and potential efficacy of iTBS in medication-free youth with the goal of supporting a future randomized controlled trial in youth with treatment-resistant major depression; 2) To assess changes in levels of psychiatric symptoms and brain imaging parameters after iTBS in youth with treatment-resistant major depression.

Endpoints:

Primary Endpoints:

Children s Depression Rating Scale (CDRS); rates of treatment completion and adverse events on standard rating scales

Secondary Endpoints:

1. Clinical Global Impression Improvement Scale (CGI-I)
2. Mood and Feelings Questionnaire (MFQ)
3. Screen for Child Anxiety Related Disorders (SCARED)
4. Resting state fMRI correlations across brain regions
5. Task-based fMRI activation to cognitive conflict
6. Fractional anisotropy on diffusion tensor imaging
7. Neurochemicals assessed by magnetic resonance spectroscopy

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Ages 13-17 at the time of enrollment
  2. Provision of signed and dated informed consent/assent form
  3. Stated willingness to comply with all study procedures and availability for the duration of the study
  4. Is considered in good health and able to fulfill all study requirements in a manner that will not adversely impact the integrity of the data, as determined by the PI after review, as applicable, of a detailed screening assessment consisting of psychiatric and medical history, mental status, physical examinations, and laboratory assessments. In some circumstances it may also be highly desirable to review medical records from healthcare providers for the 2 years prior to study enrollment, from hospitals, psychiatric facilities, and pharmacy records for the year prior to study enrollment.
  5. Youths meet DSM 5TR criteria for Major Depressive Disorder (MDD), with a current, ongoing episode of MDD being present.
  6. To enter the trial, patients must meet criteria for treatment resistance, defined in the prior study of Croarkin and coworkers as the failure to respond to adequate trials or failure to tolerate trials of at least two selective serotonin reuptake inhibitors and a trial of either cognitive behavioral therapy or Interpersonal Psychotherapy for Adolescents (IPT-A). However, to receive TMS, patients must meet criteria for a stricter definition of treatment resistance. They must fail to respond to three interventions; only subjects who received and failed all three interventions will be invited to enroll into the TMS study. This will be defined as at least 20 mg of fluoxetine, 20 mg of citalopram (or 10 mg escitalopram), and 150 mg of sertraline. One of these interventions will involve psychotherapy with either Interpersonal Psychotherapy for Adolescents (IPT-A) or cognitive behavioral therapy (CBT) for at least 12 weeks. Of note, these treatments either can be delivered in the community, as determined based on medical history, or they can be delivered as part of protocol 18-M-0037.
  7. Subject agrees to a Safety/Suicide Risk Management Protocol, which is intended to reduce the reduce the risk of suicide during study participation.
  8. Subject is currently under the care of a licensed prescriber and agrees to return to that provider upon completion of the study. During study participation, patients may continue to meet with their providers in the community, if they wish.
  9. Subject agrees, by signing Authorization for the Release of Medical Information forms (NIH-527) and informing all current providers, to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within two years of study enrollment.
  10. The participant is currently enrolled in protocol 18-M-0037

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Meets diagnostic criteria of DSM-5TR for psychosis, bipolar disorder, more than mild Autism Spectrum Disorder, ongoing severe Eating Disorder, ongoing substance use disorder (excluding nicotine) within the past month
2. In the opinion of the PI, has a current or past medical or neurological disease, condition, injury, or illness (i.e., hearing loss, increased intracranial pressure, structural brain lesion, or head trauma associated with neurological sequalae, loss of consciousness, or hospitalization) that may: (a) reduce or diminish the subject s ability to fulfill all of the study requirements; or (b) adversely affect the integrity of the data or the results of the study. This includes the need for routine use of any medication (except for contraceptive implants or oral contraceptives) for any reason.
3. Pregnancy
4. Personal history of epilepsy, seizure(s), seizure disorder, or answers Yes to any of the nine (9) questions from the epilepsy screening instrument developed by Ottman et al.
5. Has a history of, or risk factors for (history of syncope/ presyncope related to noxious stimuli, anxiety, micturition, or posture) for neurocardiogenic syncope
6. Currently receiving medication(s) that may, or is known to, reduce the seizure threshold and which, in the opinion of the PI, poses a clinically significant risk of a TMS-induced seizure that outweighs the potential benefit(s) of study participation.
7. Lifetime lack of response to an adequate trial of electroconvulsive therapy
8. Prior treatment with adequate trial of TMS
9. Vagus nerve stimulator implant or other device implants
10. Presence of intracranial implants or any other metal object within or near the head; those who have permanent retainers or other dental implants in the mouth that produce artifacts that compromise the integrity of MRI/fMRI data will be excluded from participation in this study.
11. Intellectual disability (clinically identified or IQ less than 70)
12. Symptoms of depression are due to physiologic effects of a drug of abuse or to a medical or neurological condition, as determined by the PI, based on history of contemporaneous onset of the symptoms and the associated drug or medical or neurological condition.
13. Current active suicidal ideation (i.e., presence of intent for engaging in suicidal behaviors with a plan to act on the ideation) as demonstrated by a YES response to questions 4, 5 or 6 on the Columbia-Suicide Severity Rating Scale (Screen Version - Recent). [Note: Youths with passive suicidal ideation and/or past active suicidal ideation are still eligible - Answer Yes to Questions 1, 2 or 3.]
14. Participants with recent or current history of repeated self-harm or suicide attempts occurring in the context of interpersonal conflict.
15. NIMH IRP Employees/staff and immediate family members of such staff will be excluded from the study per NIMH policy.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Treatment completion rate | End of protocol
  Rate of participants completing 20 or more iTBS sessions
Adverse event rate | Continuous
  Clinical rating on standardized scale
Clinician Depression Rating Scale | Weekly
  Clinician-rated report

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The full dataset will be shared to the extent that it is allowable by the IRB and consent process.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will work with the Clinical Director's office so that data are available six months after publication.
Access Criteria: All data will be available that are allowable based on IRB-approved procedures.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000776-M.html